CLINICAL TRIAL: NCT04333615
Title: Effects of Self-selected Walking Exercise Intensity on Adherence, Functional Capacity and Cardiovascular Risk Indicators in Patients With Peripheral Artery Disease
Brief Title: Self Selected Exercise Intensity in PAD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Raphael Mendes Ritti Dias, Professor, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SelfSelectedPAD
Record Dates: First submitted 2020-02-17; First posted 2020-04-03 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral artery disease; Exercise; Cerebral blood flow; Cardiovascular system
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Session (Sham Comparator): The control session will consist of resting on the treadmill for 30 min. It will be recommended that the patient do cycles in which he / she stands for 3 to 5 minutes and sits for 2 to 3 minutes in between, aiming to minimize the effect of body positioning on cardiovascular responses.
  Interventions: Behavioral: Exercise
- Self-selected Session (Experimental): In the self-selected exercise session, individuals will perform 30 min of exercise with self-selected intensity. This means that the duration of the series and the intensity (speed) of the treadmill are at the discretion of the patient. The important thing is that in the end it totals 30 minutes of exercise. This choice of intensity and duration of the series can be made regardless of the occurrence of pain.
  Interventions: Behavioral: Exercise
- Walking with pain (Active Comparator): In the exercise until maximum pain session (current recommendation of walking exercise prescription for patients with PAD), individuals will perform series of 3 to 5 minutes with adjusted intensity so that they feel moderate to maximum pain. This means that the patient will start walking and the Physical Education professional, experienced and able to prescribe exercises for patients with PAD, will adjust the treadmill speed so that the patient walks with moderate pain or even maximum pain. There will be rest intervals of 2 to 3 minutes. The patient will be encouraged to complete a total of 30 minutes of exercise.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Three conditions will be tested: self-selected exercise, walking with pain exercise, and control session.

SUMMARY:
Although the benefits of supervised walking training in patients with peripheral arterial disease (PAD) and symptoms of intermittent claudication (IC) are well established, one of the main problems found in this type of protocol is low adherence to training, which is possibly related to pain during training. In addition, little is known about the impact of performing exercise with pain on cerebral blood flow and cardiovascular health indicators. Thus, the objective of the present study will be to analyze the acute effects of walking exercise with self-selected intensity on the cardiovascular health indicators of patients with PAD. Therefore, 17 patients with PAD will undergo three experimental sessions: exercise with self-selected intensity, exercise until maximum pain and control. The responses of the cardiovascular variables (heart rate variability, blood pressure, heart rate, arterial stiffness and endothelial function) will be obtained before and after the sessions. In addition, during the session cardiovascular responses (cerebral blood flow, blood pressure and heart rate), perceptual and affective responses, as well as information about the exercises performed during the session will be obtained. The responses before and after exercise will be analyzed using the two-way analysis of variance for repeated measures (ANOVA) and the Newman-Keuls post-hoc test. The value of P <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral artery disease in one or both limbs (ankle brachial index <0.9);
* Claudication symptoms in six-minute walking test;
* who can walk at least 90 meters without interruption;
* that have physical conditions to perform the exercise sessions;

Exclusion Criteria:

* do not finish three experimental sessions;

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Cerebral perfusion | Change from baseline at 30 minutes after the beginning of the exercise.
  The cerebral perfusion at rest will be obtained by a transcranial doppler (TCD, Spencer Technologies, United States). To this end, patients will wear a helmet (Marc 600; Spencer Technologies, United States) capable of bilaterally attaching two 2 MHz ultrasound probes to the temporal window. With a method similar to that of an extracranial doppler, the transcranial doppler is capable of capturing the speeds of brain flows. The flow velocities of the middle cerebral artery will be measured bilaterally for 5 minutes, with patients at rest.

SECONDARY OUTCOMES:
Brachial blood pressure | Change from baseline at 30 minutes after the beginning of the exercise.
  Blood pressure will be obtained continuously by the Finometer blood pressure monitor (Finapress Medical System, Netherlands) using the beat-to-beat finger occlusion photoplethysmography technique.
Heart rate variability | Change from baseline at post-intervention, after 20 minutes.
  Heart rate variability will be assessed in order to estimate the autonomic modulation of the cardiovascular system. Therefore, after 20 minutes of rest, patients will remain in the supine position for 10 minutes, during which time RR intervals will be recorded, using a heart rate monitor valid for this function (V8000, Polar Electro, Finland).
Feeling Scale | Change from baseline at 35 minutes after the beginning of the exercise.
  A feeling scale is a single-item scale with a 11-point bipolar dimensional model, ranging from +5 to -5, commonly used to measure affective valence (pleasure / displeasure) during exercise.
Subjective perceived effort | Change from baseline at 35 minutes after the beginning of the exercise.
  The perceived effort will be evaluated using the scale adapted from subjective perception of effort (0-10 points). The perceived effort will be defined as the intensity of effort, tension and subjectively perceived fatigue that the individual feels during the exercise.
Cognitive function | Change from baseline at post-intervention, after 1 hour.
  Moca is a screening instrument were evaluating seven cognitive domains of a person and had the score between 0 and 30, where 0 is the worst score and 30 the best one. The domains will be: Visuospatial/executive functions, verbal memory, registration and learning, naming, 5-minute delayed verbal memory, attention, abstraction and orientation. A experienced researcher will explain how cognitive testes work and will apply to the patient.
Cognitive function 2 | Change from baseline at post-intervention, after 1 hour and 10 minutes.
  The Stroop test is an important tool to the assessment of the cognitive flexibility, cognitive inhibition, selective attention and information processing speed of the patient. The test consists in three phases, the first one is naming time of nonconflicting stimuli (naming colors of colored square), the second one is naming time of conflicting (where naming colors words that are printed in a different color than their meaning). The third one is to name colors of color words printed in a different color. An experienced researcher will explain how cognitive testes work and will apply to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael M Ritti Dias, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oliveira MD, Kanegusuku H, Faria DRG, Pecanha TO, Wolosker N, Correia MA, Ritti-Dias RM. Post-exercise effects of self-selected exercise intensity on cardiovascular parameters in peripheral artery disease: a randomized crossover study. Einstein (Sao Paulo). 2025 Sep 19;23:eAO1498. doi: 10.31744/einstein_journal/2025AO1498. eCollection 2025. PMID 40990702
- [Derived] de Oliveira MD, Kanegusuku H, de Faria DRG, Wolosker N, Correia MA, Ritti-Dias RM. Walking Intensity Preference of Patients With Peripheral Arterial Disease. J Cardiopulm Rehabil Prev. 2024 Jan 1;44(1):71-72. doi: 10.1097/HCR.0000000000000823. Epub 2023 Aug 30. No abstract available. PMID 37646619